CLINICAL TRIAL: NCT01643876
Title: Phase-I Clinical Trial on the Effect of Palatal Brushing on Denture Stomatitis
Brief Title: The Effect of Palatal Brushing on Denture Stomatitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Elham Emami, D.D.S., M. Sc., Ph. D, Assistant Professor, Université de Montréal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMD-UdeM-EE-2012a; NCT02201745 (obsolete NCT alias)
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Results first posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2013-12

CONDITIONS: Denture Stomatitis
Keywords: Denture stomatitis; Denture Plaque; Oral Candidiasis; Oral Hygiene
MeSH Terms: conditions — Stomatitis, Denture; Candidiasis, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Palatal brushing (Experimental): Palatal brushing after each meal for 3 months.
  Interventions: Behavioral: Palatal brushing

INTERVENTIONS:
Behavioral: Palatal brushing — Participants will be instructed to brush their palate with a manual soft-bristle brush after each meal and before sleeping for a period of 3 months. They will be asked to keep to their usual oral and denture hygiene routine during the trial to allow the isolation of the effect of palatal brushing.

SUMMARY:
Palatal brushing has several advantages including removal of debris and stimulation of blood flow and saliva, which may help to prevent or treat oral diseases, such as denture-related stomatitis in complete denture wearers.

However, there is no previous clinical trial testing this effect. Therefore, the investigators goal is to evaluate whether palatal brushing may change the severity of denture stomatitis and counts of microbes on denture and palatal mucosa.

After an initial exam and data collection, participants will receive instructions about palatal brushing and they will be assessed after 1 and 3 months. Collection of data will include patient-reported information, intraoral photographs and swabbing (for counting microbes).

Tested Hypotheses:

* There is no difference in the extent of palatal inflammation in edentulous patients with denture stomatitis before and after 3 months of palatal brushing.
* There is no difference in the number of colony forming unit (CFU) of Candida isolated from palate and denture of patients affected by denture stomatitis before and after 3 months of palatal brushing.

ELIGIBILITY:
Inclusion Criteria:

* Good general health.
* Completely edentulous maxilla.
* Currently wearing complete upper dentures.
* A clinical diagnosis of denture stomatitis.

Exclusion Criteria:

* Conditions known to promote Candida carriage such as diabetes, anemia, xerostomia, immunosuppression, chemotherapy and radiotherapy.
* Use of antibiotics, antifungal agents or corticosteroids at least 4 weeks before the study.
* Previous palatal brushing habit.
* Changing of the existing prosthesis during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elham Emami, DDS, PhD, Principal Investigator — Université de Montréal; Raphael F de Souza, DDS, PhD, Principal Investigator — University of Sao Paulo
Locations (2):
- University of Sao Paulo - Ribeirão Preto Dental School, Ribeirão Preto, São Paulo, Brazil
- Faculté de Médecine Dentaire, Université de Montréal, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from the prosthodontic clinics of the Université de Montréal and of Ribeirão Preto Dental School. Recruitment period dates: May 2012-February 2013.
Groups:
- Palatal Brushing: Palatal brushing after each meal for 3 months.
  Palatal brushing : Participants will be instructed to brush their palate with a manual soft-bristle brush after each meal and before sleeping for a period of 3 months. They will be asked to keep to their usual oral and denture hygiene routine during the trial to allow the isolation of the effect of palatal brushing.
Period: Overall Study
Arm/Group | Palatal Brushing
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Palatal Brushing
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 16
Region of Enrollment [Number; unit: participants]
  Canada | 22
  Brazil | 26

OUTCOME MEASURES:

1. Primary Outcome: Palatal Inflammation
Description: Modified Newton classification 0: Healthy mucosa
  1: Type IA, Petechiae in a normal palatal tissue, which are usually found around the orifices of the ducts of the palatal mucous glands 2: Type IB, Localized area of inflammation of the denture-bearing area 3: Type II, Generalised area of inflammation of the denture-bearing area 4: Type III, Hyperplasic palatal surface with inflammation of the denture-bearing area Inflammation area index 0: No inflammation
  1. Inflammation of the palate extending up to 25 % of the palatal denture-bearing tissue
  2. Inflammation of the palate extending between 25 % and 50 % of the palatal denture-bearing tissue
  3. Inflammation covering more than 50 % of the palatal denture-bearing tissue Inflammation severity index
  0: Normal tissue
  1. Mild inflammation
  2. Moderate inflammation
  3. Severe inflammation Total score for inflammation = area + intensity (range 0 to 6)
Time Frame: 3 months
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Palatal Brushing
Number analyzed (Participants) | 48
units on a scale
  Modified Newton classification, pre-intervention | 3 [0 to 4]
  Modified Newton classification, post-intervention | 3 [0 to 4]
  Inflammation area index, pre-intervention | 2.5 [0 to 3]
  Inflammation area index, post-intervention | 2 [0 to 3]
  Inflammation severity index, pre-intervention | 2 [0 to 3]
  Inflammation severity index, post-intervention | 1 [0 to 3]
  Total score for inflammation, pre-intervention | 5 [0 to 6]
  Total score for inflammation, post-intervention | 3 [0 to 6]
Statistical Analysis 1: Comparison: Palatal Brushing; Null hypothesis: in individuals with denture stomatitis, there are no difference in the extent of palatal inflammation before and 3 months after palatal brushing. Assuming that the minimal practically important pre/post difference in the mean change score is 20 percent and the standard deviation of the distribution of the change in score is 0.8, a sample size of 44 participants is required to ensure a power of 90 % of rejecting the null hypothesis if it is indeed false; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney); Median Difference (Net) = -1.5

2. Secondary Outcome: Candida Species Count
Description: Candida colony forming units (CFU), defined as the number of colonies formed on a 75 mm agar plate inoculated with collected samples obtained from A)plaque formed on denture surface and B)palatal mucosa.
Time Frame: 3 months
Measure: Median (Full Range); unit: colony forming units (CFUs)
Arm/Group | Palatal Brushing
Number analyzed (Participants) | 48
colony forming units (CFUs)
  Colonies from denture surface, pre-intervention | 1110 [0 to 1400000]
  Colonies from denture surface, post-intervention | 860 [0 to 380000]
  Colonies from palatal mucosa, pre-intervention | 0 [0 to 3440]
  Colonies from palatal mucosa, post-intervention | 0 [0 to 2560]
Statistical Analysis 1: Comparison: Palatal Brushing; Null Hypothesis: in individuals with denture stomatitis, there are no difference in the number of Candida Colony-Forming Units (CFUs), before and 3 months after palatal brushing; Test type: Superiority or Other; p < 0.05, Wilcoxon (Mann-Whitney); Median Difference (Net) = -57.5

ADVERSE EVENTS:
Time Frame: 3 months.
Description: 48 participants were assessed for adverse events. "0"Participants had any serious and/or non-serious adverse events after 3 months of assessment.
Arm/Group | Palatal Brushing
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

LIMITATIONS AND CAVEATS:
One group pre-test post-test study. External validity limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes